CLINICAL TRIAL: NCT02165618
Title: Rationalisation of Polypharmacy by the Geriatric Consultation Team Using the RASP List: a Pilot Study
Brief Title: Rationalisation of Polypharmacy by the Geriatric Consultation Team
Acronym: RASP-GCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: S-54896
Record Dates: First submitted 2014-05-26; First posted 2014-06-17 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-05

CONDITIONS: Iatrogenic Disease
Keywords: frailty; geriatric, elderly; polypharmacy
MeSH Terms: conditions — Iatrogenic Disease; Frailty | interventions — Medication Review

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GCT (No Intervention): In a before phase, data on how the GCT operated (i.e. good clinical practice) was gathered.
- GCT-RASP (Active Comparator): Medication review, based on but not limited to the RASP list
  Interventions: Other: Medication review, based on but not limited to the RASP list

INTERVENTIONS:
Other: Medication review, based on but not limited to the RASP list — Systematic approach:
  1. Medication reconciliation
  2. Applying the RASP list
  3. Expert review (not based on the RASP list)
  4. Multidisciplinary discussion
  Other Names: RASP; RASP list; Systematic medication review
  Arms: GCT-RASP

SUMMARY:
Polypharmacy is a common problem in elderly, leading among others to increased adverse drug events. The aim of this pilot study was to evaluate whether a systematic medication evaluation by a geriatric consultation team using the RASP (Rationalisation of drugs on admission by an adjusted STOPP*-list in older patients) list could reduce inappropriate prescribing for elderly admitted patients, admitted to non-geriatric departments.

(* = Screening Tool of Older Persons' potentially inappropriate Prescriptions)

DETAILED DESCRIPTION:
Polypharmacy and (potentially) inappropriate prescribing is highly prevalent in the older population, associated with increase health care expenditures, morbidity and avoidable adverse events .

The aim of this pilot study was to evaluate whether a systematic medication evaluation by a geriatric consultation team (GCT) using the RASP (Rationalisation of drugs on admission by an adjusted STOPP-list in older patients) list could reduce inappropriate prescribing for older admitted patients, admitted to non-geriatric departments. The GCT could offer the ideal format to deliver the intervention to a broad older hospitalised population.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to a non-geriatric ward
* 75 years or older
* Dutch speaking
* Consultation by the GCT

Exclusion Criteria:

* End-of-life
* No drugs on admission

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Number of medication-related recommendations by the geriatric consultation team. | The number was ascertained at time of discharge from the ward, taking into account an average hospital stay of 14 days.

SECONDARY OUTCOMES:
Number of potentially inappropriate drugs at discharge, as identified by the RASP list. | The number was ascertained at time of discharge from the ward, taking into account an average hospital stay of 14 days.
Number of drugs at discharge, relative to the drugs on admission. | The number was ascertained at time of discharge from the ward, taking into account an average hospital stay of 14 days.
Acceptance rate of the GCT interventions by the treating physician. | Up to 72 hours after the GCT had given its recommendations.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenz R Van der Linden, PharmD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Johan Flamaing, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Jos Tournoy, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Flemish Brabant, Belgium

REFERENCES:
- [Derived] Van der Linden L, Hias J, Dreessen L, Milisen K, Flamaing J, Spriet I, Tournoy J. Medication review versus usual care to improve drug therapies in older inpatients not admitted to geriatric wards: a quasi-experimental study (RASP-IGCT). BMC Geriatr. 2018 Jul 3;18(1):155. doi: 10.1186/s12877-018-0843-y. PMID 29970005